CLINICAL TRIAL: NCT05181618
Title: A Multicenter, Open-Label Phase IV Study to Evaluate Overall Health, Physical Activity, and Joint Outcomes, in Participants Aged ≥13 and <70 Years With Severe or Moderate Hemophilia A Without FVIII Inhibitors on Emicizumab Prophylaxis
Brief Title: A Study to Evaluate Overall Health, Physical Activity, and Joint Outcomes in Participants With Severe or Moderate Hemophilia A Without Factor VIII Inhibitors on Emicizumab Prophylaxis
Acronym: Beyond ABR
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MO42623; 2020-005092-13 (EudraCT Number); 2023-505747-40-00 (Registry Identifier: EU CT Number); ISRCTN10101701 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2021-12-06; First posted 2022-01-06 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Severe Hemophilia A; Moderate Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — emicizumab

STUDY DESIGN:
Intervention Model Description: The intervention study model is "single group" because all three cohorts of participants with hemophilia A will be receiving the same intervention: emicizumab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1, Hemophilia A and Without Arthropathy: Emicizumab (Experimental): Cohort 1 comprises participants with severe or moderate hemophilia A and with no synovitis and no osteochondral damage (Haemophilia Early Arthropathy Detection with Ultrasound [HEAD-US] score of 0) in all index joints.
  Interventions: Drug: Emicizumab
- Cohort 2, Hemophilia A and with Synovitis Only: Emicizumab (Experimental): Cohort 2 comprises participants with severe or moderate hemophilia A and with synovitis (HEAD-US synovitis score of ≥1) in at least one index joint and no osteochondral damage (HEAD-US bone and cartilage score of 0).
  Interventions: Drug: Emicizumab
- Cohort 3, Hemophilia A and with Osteochondral Damage: Emicizumab (Experimental): Cohort 3 comprises participants with severe or moderate hemophilia A and with osteochondral damage (HEAD-US bone and cartilage score of ≥1) in at least one index joint and with any synovitis score.
  Interventions: Drug: Emicizumab

INTERVENTIONS:
Drug: Emicizumab — The emicizumab dosing regimen will be 3 milligrams per kilogram of body weight (mg/kg) subcutaneously (SC) once a week (QW) for 4 weeks followed by participant preference of one of the following maintenance regimens: 1.5 mg/kg QW, 3 mg/kg once every 2 weeks (Q2W), or 6 mg/kg once every 4 weeks (Q4W) in agreement with the investigator.
  Other Names: Hemlibra; RO5534262; RG6013; ACE910

SUMMARY:
Study MO42623 is a Phase IV, multicenter, open-label, three cohort study designed to evaluate the impact of emicizumab prophylaxis on overall health, physical activity, and joint outcomes in participants aged ≥13 and <70 years with severe hemophilia A without factor VIII (FVIII) inhibitors or moderate hemophilia A without FVIII inhibitors who are receiving FVIII prophylaxis and who will start emicizumab treatment as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe congenital hemophilia A (intrinsic factor VIII [FVIII] level <1%) or moderate congenital hemophilia A (intrinsic FVIII level ≤5%) if previously prescribed prophylaxis
* A negative test for FVIII inhibitor (i.e., <0.6 Bethesda Units) during screening period
* No history of FVIII inhibitory antibodies (<0.6 BU/mL using the Bethesda assay) in the last 5 years. Participants who completed successful immune tolerance induction (ITI) at least 5 years before screening are eligible, provided they have had no evidence of inhibitor recurrence (permanent or temporary) as may be indicated by detection of an inhibitor, FVIII half-life <6 hours, or FVIII recovery <66% since completing ITI
* Participants who were on standard FVIII prophylaxis, defined as the regular administration of FVIII to prevent bleeding, for at least the last 24 weeks, can be enrolled regardless of the number of bleeds during this period
* Adequate hematologic, hepatic and renal function
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception during the treatment period and for at least 24 weeks after the final dose of emicizumab

Exclusion Criteria:

* Inherited or acquired bleeding disorder other than severe congenital hemophilia A (intrinsic FVIII level <1%) or moderate congenital hemophilia A (intrinsic FVIII level ≤5%) without FVIII inhibitors who were previously prescribed prophylaxis for at least 24 weeks
* Participants who have previously received emicizumab prophylaxis
* Participants that plan to have joint replacement, joint procedure, synovectomy or synoviorthesis at screening
* Participants who had joint replacement, joint procedure, synovectomy or synoviorthesis: Less than 2 years ago; OR, More than 3 years ago and are still experiencing pain in the joint. For participants who had joint replacement, joint procedure, synovectomy or synoviorthesis more than 2 years ago who are not experiencing pain in the joint(s), the participant may be enrolled but the specific joint(s) in which the procedure was conducted will be excluded from the study
* Participants who have conditions other than hemophilia A that can affect joint health and structure (e.g., osteoarthritis) or with severely impaired mobility due to conditions other than hemophilia A
* Participants with known reduced bone mineral density defined as clinically relevant vitamin D deficiency
* Participants with pre-existing uncontrolled or unstable cardiovascular disease not receiving targeted medication or in a stable condition
* Participants not eligible for MRI
* History of illicit drug or alcohol abuse within 48 weeks prior to screening in the investigator's judgement
* Participants who are at high risk for thrombotic microangiopathy (TMA)
* Previous (within the last 12 months) or current treatment for thromboembolic disease (with the exception of previous catheter-associated thrombosis for which anti-thrombotic treatment is not currently ongoing) or signs of thromboembolic disease
* Other conditions (e.g., certain autoimmune diseases) that may currently increase the risk of bleeding or thrombosis
* History of clinically significant hypersensitivity associated with monoclonal antibody therapies or components of the emicizumab injection
* Planned surgery during the emicizumab loading dose phase
* Known HIV infection not controlled by medication
* Concomitant disease, condition, significant abnormality on screening evaluation or laboratory tests, or treatment that could interfere with the conduct of the study, or that would in the opinion of the investigator, pose an additional unacceptable risk in administering study drug to the participant
* Receipt of any of the following: An investigational drug to treat or reduce the risk of hemophilic bleeds within 5 half-lives of last drug administration at screening; A non-hemophilia-related investigational drug within last 30 days or 5 half-lives at screening, whichever is shorter; or, Any other investigational drug currently being administered or planned to be administered
* Inability to comply with the study protocol
* Pregnant or breastfeeding, or intending to become pregnant during the study

Ages: 13 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2026-12-04 (Estimated); Study Completion 2027-05-21 (Estimated)

PRIMARY OUTCOMES:
Joint Status at 6 Months, Based on Centrally Reviewed Haemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) Scores with a Specific Focus on the Synovitis Score in Participants with Synovitis | 6 Months
Joint Status at 12 Months, Based on Centrally Reviewed Haemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) Scores with a Specific Focus on the Synovitis Score in Participants with Synovitis | 12 Months
Joint Status at 24 Months, Based on Centrally Reviewed Haemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) Scores with a Specific Focus on the Synovitis Score in Participants with Synovitis | 24 Months
Joint Status at 36 Months, Based on Centrally Reviewed Haemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) Scores with a Specific Focus on the Synovitis Score in Participants with Synovitis | 36 Months
Clinical Joint Status at 6 Months, Based on the Hemophilia Joint Health Score (HJHS v2.1) Excluding Gait Assessment | 6 Months
Clinical Joint Status at 12 Months, Based on the Hemophilia Joint Health Score (HJHS v2.1) Excluding Gait Assessment | 12 Months
Clinical Joint Status at 24 Months, Based on the Hemophilia Joint Health Score (HJHS v2.1) Excluding Gait Assessment | 24 Months
Clinical Joint Status at 36 Months, Based on the Hemophilia Joint Health Score (HJHS v2.1) Excluding Gait Assessment | 36 Months
Joint Status at 36 Months, Based on Centrally Reviewed International Prophylaxis Study Group (IPSG) Score (with MRI) | 36 Months
Number of Problem Joints at 6 Months | 6 Months
  Problem joints are defined as joints having chronic joint pain and/or limited range of movement due to compromised joint integrity (i.e., chronic synovitis and/or hemophilic arthropathy) with or without persistent bleeding.
Number of Problem Joints at 12 Months | 12 Months
  Problem joints are defined as joints having chronic joint pain and/or limited range of movement due to compromised joint integrity (i.e., chronic synovitis and/or hemophilic arthropathy) with or without persistent bleeding.
Number of Problem Joints at 24 Months | 24 Months
  Problem joints are defined as joints having chronic joint pain and/or limited range of movement due to compromised joint integrity (i.e., chronic synovitis and/or hemophilic arthropathy) with or without persistent bleeding.
Number of Problem Joints at 36 Months | 36 Months
  Problem joints are defined as joints having chronic joint pain and/or limited range of movement due to compromised joint integrity (i.e., chronic synovitis and/or hemophilic arthropathy) with or without persistent bleeding.
Percentage of Joints That are Problem Joints at 6 Months | 6 Months
Percentage of Joints That are Problem Joints at 12 Months | 12 Months
Percentage of Joints That are Problem Joints at 24 Months | 24 Months
Percentage of Joints That are Problem Joints at 36 Months | 36 Months
Change from Baseline in the CATCH Domain Scores Over Time, as Assessed with the Comprehensive Assessment Tool of Challenges in Hemophilia (CATCH) Questionnaire for Adult Participants | At Baseline (Day 1), Months 3, 6, 9, 12, 18, 24, 30, and 36
Change from Baseline in the CATCH Domain Scores Over Time, as Assessed with the CATCH Questionnaire for Pediatric Participants | At Baseline (Day 1), Months 3, 6, 9, 12, 18, 24, 30, and 36
Change from Baseline in the Average Daily Time Spent Doing Physical Activities by Intensity Level Over Time, as Assessed by Participant Responses to the International Physical Activity Questionnaire Short Format (IPAQ-SF) | At Baseline (Day 1), Months 3, 6, 9, 12, 18, 24, 30, and 36
Daily Step Count Over Time, as Measured with a Wearable Activity Tracker | From Baseline until end of treatment period (up to 36 months)
Daily Metabolic Equivalents of Tasks (METs) Over Time, as Measured with a Wearable Activity Tracker | From Baseline until end of treatment period (up to 36 months)
Daily Time Spent in Moderate to Vigorous Physical Activity (MVPA) Over Time, as per the Activity Tracker Default Categorization | From Baseline until end of treatment period (up to 36 months)
Daily Active Minutes of Physical Activity Over Time, as Measured with a Wearable Activity Tracker | From Baseline until end of treatment period (up to 36 months)
Model-Based Annualized Bleed Rates for All Bleeds, Treated Bleeds, Spontaneous Bleeds, Joint Bleeds, Treated Joint Bleeds, and Target Joint Bleeds | From Baseline until end of treatment period (up to 36 months)
Mean Calculated Annualized Bleed Rates for All Bleeds, Treated Bleeds, Spontaneous Bleeds, Joint Bleeds, Treated Joint Bleeds, and Target Joint Bleeds | From Baseline until end of treatment period (up to 36 months)
Median Calculated Annualized Bleed Rates for All Bleeds, Treated Bleeds, Spontaneous Bleeds, Joint Bleeds, Treated Joint Bleeds, and Target Joint Bleeds | From Baseline until end of treatment period (up to 36 months)
Number of Participants who Prefer Emicizumab SC Treatment, Their Previous Hemophilia IV Treatment, or Have No Preference, as Assessed Through Use of the Emicizumab Preference Survey at Month 6 | At Month 6

SECONDARY OUTCOMES:
Number of Participants with at Least One Adverse Event, with Severity Determined According to the World Health Organization (WHO) Toxicity Scale | From Baseline until 24 weeks after the final dose of emicizumab (up to 3.5 years)
Number of Participants with at Least One Thromboembolic Event | From Baseline until 24 weeks after the final dose of emicizumab (up to 3.5 years)
Number of Participants with at Least One Event of Thrombotic Microangiopathy (TMA) | From Baseline until 24 weeks after the final dose of emicizumab (up to 3.5 years)
Number of Participants with at Least One Severe Hypersensitivity, Anaphylaxis, and Anaphylactoid Event | From Baseline until 24 weeks after the final dose of emicizumab (up to 3.5 years)
Number of Participants with at Least One Injection-Site Reaction | From Baseline until 24 weeks after the final dose of emicizumab (up to 3.5 years)
Number of Participants with Anti-Drug Antibodies (ADAs) Against Emicizumab at Baseline and During the Study | At Baseline, Months 6, 12, 24, and 36
Number of Participants who Develop Anti-FVIII Inhibitors During the Study | At Months 6, 12, 24, and 36

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (28):
- United States (3):
  - Orthopaedic Institute for Children, Los Angeles, California
  - University of Miami Medical Center, Miami, Florida
  - Oklahoma Children's Hospital ? Jimmy Everest Center, Oklahoma City, Oklahoma
- Brazil (2):
  - Hospital das Clinicas - UNICAMP, Campinas, São Paulo
  - Hospital das Clínicas Faculdades Médicas de Ribeirão Preto, Ribeirão Preto, São Paulo
- Hamilton Health Sciences Corporation, Hamilton, Ontario, Canada
- Germany (2):
  - Charité Universitätsklinikum Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
- Észak-Pesti Centrumkórház - Honvédkórház, Budapest, Hungary
- Italy (4):
  - AOU Federico II, Napoli, Campania
  - Policlinico Univ. A. Gemelli, Rome, Lazio
  - IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - AOU Careggi, Florence, Tuscany
- Hôpital d'enfants de Rabat - Service d'hémato-oncologie pédiatrique, Rabat, Morocco
- University Clinical Centre of Serbia, Belgrade, Serbia
- Spain (5):
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall de Hebron, Barcelona
  - Hospital Universitario la Paz, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
- Tunisia (2):
  - CHU Farhat Hached, Sousse
  - Aziza Othmana Hospital, Tunis
- Turkey (Türkiye) (4):
  - Gazi Universitesi Tip Fakultesi, Ankara
  - Akdeniz Uni School of Medicine, Antalya
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Ege Uni Medical School, Izmir
- United Kingdom (2):
  - St Thomas Westminster, London
  - Manchester University NHS Foundation Trust (MFT), Manchester

IPD SHARING:
Plan to Share IPD: No